CLINICAL TRIAL: NCT02934464
Title: Assessment of Ramucirumab Plus Paclitaxel as Switch MANteInance Versus Continuation of First-line Chemotherapy in Patients With Advanced HER-2 Negative Gastric or Gastroesophageal Junction Cancers: the ARMANI Phase III Trial
Brief Title: Assessment of Ramucirumab Plus Paclitaxel as Switch MANteInance Versus Continuation of First-line Chemotherapy in Patients With Advanced HER-2 Negative Gastric or Gastroesophageal Junction Cancers
Acronym: ARMANI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT 103-16
Record Dates: First submitted 2016-10-06; First posted 2016-10-17 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ramucirumab; Paclitaxel; Oxaliplatin; Leucovorin; XELOX; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Experimental): * RAMUCIRUMAB 8 mg/kg on Days 1 and 15 of every 28-day cycle
  * PACLITAXEL 80 mg/m2 on Days 1, 8, and 15 of every 28-day cycle until progressive disease, unacceptable toxicity, informed consent withdrawal or patient's death.
  Interventions: Drug: RAMUCIRUMAB; Drug: Paclitaxel
- ARM B (Active Comparator): * FOLFOX4: Oxaliplatin 85 mg/m2 + l-Leucovorin 100 mg/m2 + 5-fluorouracil 400/600 mg/m2. Cycle length is 2 weeks +/- 3 days.
  * mFOLFOX6: Oxaliplatin a 85 mg/m2+ l-Leucovorin 200 mg/m2 + 5-fluorouracil 400 mg/m2 and 2400 mg/m2 46-hours continous infusion. Cycle length is 2 weeks +/- 3 days.
  * XELOX:Oxaliplatin130 mg/m2 + Capecitabine will be 2000 mg/m2 for 14 days. Cycle length is 3 weeks +/- 3 days.
  Interventions: Drug: FOLFOX 4; Drug: mFOLFOX 6; Drug: XELOX

INTERVENTIONS:
Drug: RAMUCIRUMAB
  Other Names: Cyramza
  Arms: ARM A
Drug: Paclitaxel — Paclitaxel
  Arms: ARM A
Drug: FOLFOX 4
  Other Names: Oxaliplatino + l-leucovorin + 5 Fluorouracile
  Arms: ARM B
Drug: mFOLFOX 6
  Other Names: Oxaliplatino + l-leucovorin + 5 Fluorouracile
  Arms: ARM B
Drug: XELOX
  Other Names: Oxaliplatino + Capecitabina
  Arms: ARM B

SUMMARY:
This is a randomized, open-label, multicenter phase III trial of ramucirumab plus paclitaxel, given as switch maintenance, versus continuation of first-line chemotherapy, given as per standard clinical practice, in subjects with unresectable locally advanced or metastatic HER-2 negative gastric or GEJ cancer, without disease progression following 3 months of first-line doublet chemotherapy.

The acceptable first-line or lead-in chemotherapy will be:

* FOLFOX4:Oxaliplatin 85 mg/m2. l-Leucovorin 100 mg/m2 5-fluorouracil 400/600 mg/m2. Cycle length is 2 weeks +/- 3 days.
* ModifiedFOLFOX6: Oxaliplatin a 85 mg/m2. l-Leucovorin 200 mg/m2. 5-fluorouracil 400 mg/m2 and 2400 mg/m2 46-hours continous infusion. Cycle length is 2 weeks +/- 3 days.
* XELOX:Oxaliplatin130 mg/m2.Capecitabine will be 2000 mg/m2 for 14 days. Cycle length is 3 weeks +/- 3 days.

DETAILED DESCRIPTION:
Treatment must be continued for up to 4 three-weekly cycles or 6 bi-weekly cycles, or for up to a maximum of 12 weeks. Subjects with CR/PR/SD after oxaliplatinum compound and fluoropyrimidine-based regimens, or without evidence of progressive disease in case of non-measurable disease, will be randomized in 1:1 ratio between the two treatment arms.

Prior to randomization, subjects will be stratified based on Center; Prior gastrectomy: No vs. Yes; Peritoneal carcinomatosis: Yes vs. No; Site of origin: GEJ vs. gastric.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

1. Written informed consent prior to performance of any study procedure;
2. Age ≥18 years;
3. ECOG Performance Status 0-1 (Appendix I);
4. Life expectancy of at least 12 weeks in the opinion of the Investigator;
5. Unresectable locally advanced or metastatic, histopathologically confirmed, HER-2 negative adenocarcinoma of gastric or GEJ cancer with measurable and/or evaluable disease based on RECIST, v1.1
6. Must have received lead-in chemotherapy in the first-line setting using one of the fluoropyrimidines- and oxaliplatin-based doublet combinations as specified in Section 7 and continued for three months (i.e. 6 administrations for bi-weekly cycles regimens or 4 administrations for three-weekly cycles regimens). Patients who had received adjuvant cisplatin/oxaliplatin plus fluoropyrimidine-based doublet chemotherapy and had recurrence beyond 12 months from its completion are eligible.
7. Must have radiological evidence of clinical benefit following the last dose of the lead-in chemotherapy (either CR, PR or SD by RECIST v1.1 criteria in case of measurable disease, or absence of progressive disease in case of non-measurable disease).
8. Laboratory requirements:

   * The patient has adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥1000/µL, hemoglobin ≥9 g/dL (5.58 mmol/L), and platelets ≥100,000/µL.
   * The patient has adequate hepatic function as defined by a total bilirubin ≤1.5 mg/dL (25.65 μmol/L), and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 times the upper limit of normal (ULN; or 5.0 times the ULN in the setting of liver metastases).
   * The patient has adequate renal function as defined by a serum creatinine ≤1.5 times the ULN, or creatinine clearance (measured via 24-hour urine collection) ≥40 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed). The patient's urinary protein is ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol).
   * Coagulation: The patient must have adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Patients receiving warfarin must be switched to low molecular weight heparin and have achieved stable coagulation profile prior to randomization
9. Patients must be accessible for treatment and follow up. Patients registered on this trial must be treated and followed at the participating center.
10. Archival tumor tissue is required for exploratory research at enrollment.
11. Because the teratogenicity of ramucirumab is not known, the patient, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods) for the entire duration of the study including a minimum of 12 weeks after dosing has been completed. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrolment. Women must not be breastfeeding.

Exclusion Criteria:

Exclude a patient from this study if any of the following conditions are observed:

1. HER2 positive status, or the patient has squamous cell.
2. Prior malignancy, active within 3 years from study entry, except for locally curable cancers that have been apparently cured and need no subsequent therapy, such as non-melanoma skin cancers, superficial bladder cancer or cancer in situ of the breast or cervix.
3. Has a serious illness or medical condition(s) including, but not limited to the following:

   1. Known brain metastasis or leptomeningeal metastasis.
   2. Active infection (ie, body temperature ≥38°C due to infection).
   3. Ascites, pleural effusion or pericardial fluid requiring drainage in last 4 weeks.
   4. Intestinal obstruction, pulmonary fibrosis or interstitial pneumonitis, renal failure, liver failure, or cerebrovascular disorder.
   5. Uncontrolled diabetes.
   6. The patient has symptomatic congestive heart failure (New York Heart Association II-IV) or symptomatic or poorly controlled cardiac arrhythmia.
   7. The patient has experienced any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to randomization.
   8. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or hepatitis B or C.
   9. Autoimmune disorders or history of organ transplantation that require immunosuppressive therapy.

   l.Psychiatric disease that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results.

   m.The patient has a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to randomization.

   n.The patient is receiving therapeutic anticoagulation with warfarin, low-molecular weight heparin or similar agents. Patients receiving prophylactic, low-dose anticoagulation therapy are eligible provided that the coagulation parameters defined in the inclusion criteria (INR ≤ 1.5 and aPTT ≤ 1.5 x ULN) or (PT ≤ 1.5 x ULN and aPTT ≤1.5 x ULN) are met.

   o.The patient is receiving chronic therapy with nonsteroidal anti-inflammatory agents (NSAIDs, eg, indomethacin, ibuprofen, naproxen or similar agents) or other anti-platelet agents (eg, clopidogrel, ticlopidine, dipyridamole, anagrelide). Aspirin use at doses up to 325 mg/day is permitted.

   p.The patient has significant bleeding disorders, vasculitis, or had a significant bleeding episode from the gastrointestinal tract within 3 months prior to study entry.

   q.History of gastrointestinal perforation and/or fistulae within 6 months prior randomization.

   r.The patient has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.

   s.The patient has uncontrolled arterial hypertension ≥ 150 / ≥ 90 mm Hg despite standard medical management.

   t.The patient has a serious or non healing wound or peptic ulcer or bone fracture within 28 days prior to randomization.

   u.Known allergy or hypersensitivity to monoclonal antibody treatment or any components used in the ramucirumab DP preparation. Known allergy or hypersensitivity to paclitaxel or any components used in the paclitaxel preparation or other contraindication for taxane therapy.

   v.Persistent proteinuria of CTCAE Grade 3 (>3.5g/24 hours).
4. Treatment with any of the following within the specified time frame prior to study drug administration:

   1. Major surgery within 28 days prior to randomization, or central venous access device placement within 7 days prior to randomization.
   2. Any investigational agent including VEGF or VEGFR-targeted agents within prior 4 weeks
   3. Extended field radiation within prior 4 weeks or limited field radiation within prior 2 weeks.
5. Unresolved toxicity of greater than or equal to CTCAE Grade 2 attributed to any prior therapies (excluding anemia, alopecia, skin pigmentation). In particular, patients with platinum induced neurotoxicity greater than or equal CTCAE Grade 2 that has not resolved after induction phase should be excluded.
6. Is a pregnant or lactating female, or is planning to become pregnant during treatment and within 12 weeks after the end of treatment with ramucirumab. Women of child-bearing potential with either positive or no pregnancy test at baseline. Women of child-bearing potential or sexually active men not willing to use contraception during study and for at least 12 weeks after end of treatment with ramucirumab. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-child bearing potential.
7. Concomitant participation or participation within the last 30 days in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 3 years
  Progression-Free Survival (PFS)

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Overall Survival (OS)
Time-to-treatment failure | 3 years
  Time-to-treatment failure
Overall response rate | 3 years
  Overall response rate
Duration of response | 3 years
  Duration of response of patients who receive swich maintenance (arm A) versus patients who receive continuation therapy (arm B).
Percentage of patients in second line therapy | 3 years
  To compare the percentage of patients that will receive a second line therapy according to arm treatment.
Adverse events | 3 years
  Incidence of adverse events, according to CTCAE v4.03
Quality of life EORTC QLQ-C30 | 3 years
  PRO are assessed using the questionnaires EORTC QLQ-C30
Quality of life EORTC QLQ-OG25 | 3 years
  PRO are assessed using the questionnaire the EORTC QLQ-OG25
Quality of life EuroQol EQ-5D | 3 years
  PRO are assessed using the questionnaire EuroQol EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: MARIA DI BARTOLOMEO, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (1):
- Maria Di Bartolomeo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Randon G, Lonardi S, Fassan M, Palermo F, Tamberi S, Giommoni E, Ceccon C, Di Donato S, Fornaro L, Brunetti O, De Vita F, Bittoni A, Chini C, Spallanzani A, Nappo F, Bethaz V, Strippoli A, Latiano T, Cardellino GG, Giuliani F, Morano F, Niger M, Raimondi A, Prisciandaro M, Pircher CC, Sciortino C, Marchesi S, Garattini SK, Airo G, Miceli R, Di Bartolomeo M, Pietrantonio F. Ramucirumab plus paclitaxel as switch maintenance versus continuation of first-line oxaliplatin-based chemotherapy in patients with advanced HER2-negative gastric or gastro-oesophageal junction cancer (ARMANI): a randomised, open-label, multicentre, phase 3 trial. Lancet Oncol. 2024 Dec;25(12):1539-1550. doi: 10.1016/S1470-2045(24)00580-1. Epub 2024 Nov 15. PMID 39557058
- [Derived] Di Bartolomeo M, Niger M, Morano F, Corallo S, Antista M, Tamberi S, Lonardi S, Di Donato S, Berardi R, Scartozzi M, Cardellino GG, Di Costanzo F, Rimassa L, Luporini AG, Longarini R, Zaniboni A, Bertolini A, Tomasello G, Pinotti G, Scagliotti G, Tortora G, Bonetti A, Spallanzani A, Frassineti GL, Tassinari D, Giuliani F, Cinieri S, Maiello E, Verusio C, Bracarda S, Catalano V, Basso M, Ciuffreda L, De Vita F, Parra HS, Fornaro L, Caporale M, de Braud F, Pietrantonio F. Assessment of Ramucirumab plus paclitaxel as switch maintenance versus continuation of first-line chemotherapy in patients with advanced HER-2 negative gastric or gastroesophageal junction cancers: the ARMANI phase III trial. BMC Cancer. 2019 Mar 29;19(1):283. doi: 10.1186/s12885-019-5498-3. PMID 30922323